CLINICAL TRIAL: NCT02075138
Title: An Observational Multi-Centre Field Study to Assess Symptom Scores and Allergy Medication Usage in Subjects With a History of Grass-Induced Rhinoconjunctivitis
Brief Title: Grass Observational Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Syneos Health (Other); CIDAL (Unknown)
Responsible Party: Sponsor
Other Study IDs: TG003
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Grass Allergy; Rhinoconjunctivitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Grass-Induced Rhinoconjunctivitis Subjects

SUMMARY:
Grass pollen allergens are universally recognised as a major cause of allergic diseases in humans, including asthma, allergic rhinitis, conjunctivitis and dermatitis.

The purpose of the current study is to evaluate allergy symptoms and allergy medication in subjects with grass-related rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* History of moderate to severe rhinoconjunctivitis consistent with allergy to grass for at least 2 years.
* Forced Expiratory Volume in 1 Second (FEV1) of at least 70% of predicted value or personal best if available at the Screening Visit.
* Perennial Rye grass or Timothy grass-specific IgE ≥ 0.35 kU/L as measured by ImmunoCAP®.
* Positive skin prick test to Perennial Rye grass or Timothy grass allergen

Exclusion Criteria:

* Positive skin prick test ≥ 5 mm to any confounding, co-existing seasonal allergens likely to be present during the pre-season baseline and grass pollen period.
* Medical records of symptomatic perennial allergic rhinitis and/or asthma or a positive skin test ≥ 5 mm due to a perennial allergen to which the subject is regularly exposed (moulds, dust mites, cockroaches, and animal dander) and which cannot be avoided during the course of the study.
* Previous immunotherapy treatment with any grass allergen for more than 1 month within 5 years prior to screening.
* Subjects who had been treated with any non-grass licensed allergen immunotherapy extracts or non-grass investigational immunotherapy for more than 1 month within 1 year.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a history of Grass induced Rhinoconjunctivitis
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To evaluate Total Rhinoconjunctivitis Symptom Score and allergy medication use as a combine score | 6 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Washington D.C., District of Columbia
  - Normal, Illinois
  - Sylvania, Ohio
  - Medford, Oregon
  - Spokane, Washington
- Buenos Aires City, Buenos Aires, Argentina
- Temuco, Región de la Araucanía, Chile